CLINICAL TRIAL: NCT04372160
Title: Cross-sectional Study to Assess the Extent of Agreement Between an Online 24-hr Dietary Recall and an Interviewer-administered 24-hr Dietary Recall on the Same Day for 2 Non-consecutive Days 1 wk Apart to Adults and School Age Children in Order to Compare Energy and Nutrient Intakes Derived From the Two Methods and Conduct User Evaluation of the Online Dietary Assessment Tool
Brief Title: Assess Extent of Agreement Between Online 24-hr Dietary Recall and Interviewer-administered 24-hr Dietary Recall on the Same Day for 2 Non-consecutive 2 Days 1 wk Apart to Adults and School Age Children
Status: Completed | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-1803
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Dietary Habits
Keywords: 24-hr dietary recall
MeSH Terms: conditions — Feeding Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Younger school age children: Equal ratio of boys and girls, age range 7-13 years (68 subjects)
  Interventions: Other: Dietary assessment
- Older school age children: Equal ratio of boys and girls), age range 14-17 years (68 subjects)
  Interventions: Other: Dietary assessment
- Adults: Equal ratio of adult men and women, age range 18-65 years (68 subjects).
  Interventions: Other: Dietary assessment

INTERVENTIONS:
Other: Dietary assessment — 24-hr dietary recall

SUMMARY:
Hypothesis: The online 24 hour dietary recall will be comparable to interviewer-administered 24 hour dietary recall considering the limits of agreement in the reporting of energy and macronutrient intake. If the two methods of dietary assessment are comparable (i.e., if greater than 95% of the data plots will lie within the limits of agreement), the online dietary assessment tool could be used in future studies to collect dietary intake data and health data in larger sets of Russian populations, in order to investigate the potential differences in anthropometric risk factors of non-communicable diseases (cancers, diabetes, obesity, hypertension, mortality, etc.) in people with different diet.

DETAILED DESCRIPTION:
Baseline assessments include a demographic questionnaire, including anthropometrics (height, weight), a heath status questionnaire, supplement intake, eating habits, and a food frequency questionnaire, and cardiovascular assessment (blood pressure and heart rate).

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be male and female.
2. 7-65 years of age.
3. Must be willing and able to record (via online questionnaire) the prior day's food intake according to the protocol.
4. Understanding of the procedures to be undertaken as part of the study.
5. Willingness to participate in research measurement and follow instructions provided by the investigator.
6. Informed, voluntary, written consent to participate in the study.

Exclusion Criteria:

1. Currently have any disease or condition that required chronic therapeutic nutritional treatment (the use of specific nutrition services to treat an illness, injury, or condition).
2. Currently dieting (currently on a diet to lose weight; currently on a diet for health reasons; currently on a diet to gain weight).
3. Have any formal training in nutrition, or had prior experience completing dietary recalls.
4. Participant is unable to complete computer-based dietary questionnaires, through a mental, physical or visual limitation that would preclude him/her from reporting their dietary intake.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recruited at 3 locations within a specific area: Saint-Petersbourg Russia
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Extent of agreement between online self-administered online 24 hour dietary recall and interviewer-administered 24 hour dietary recall in energy and nutrient reporting | The average of the two 24 hour periods (recall 1 and recall 2) within each method. Recall 1 and Recall 2 are in-person visits one week apart.
  Bland Altman analysis of energy and macronutrient (carbohydrates, fat, protein) intake. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately.

SECONDARY OUTCOMES:
Difference between the self-administered online 24 hour dietary recall and the interviewer-administered 24 hour dietary recall in the reporting of energy and nutrient intake. | The average of the two 24 hour periods (recall 1 and recall 2) within each method. Recall 1 and Recall 2 are in-person visits one week apart.
  Absolute and percent difference. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately.
Correlation between estimates of energy and nutrient intake reported by self-administered online 24 hour dietary recall and the interviewer-administered 24 hour dietary recall for the same day. | The average of the two 24 hour periods (recall 1 and recall 2) within each method. Recall 1 and Recall 2 are in-person visits one week apart.
  Cross-classification analysis. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately. The relative agreement will be in quartiles: exact agreement, exact plus adjacent quartile, disagreement or extreme disagreement.
Extent of agreement between measured and self-reported body mass index (BMI) | The average body mass index (BMI) in kg/m squared of the two 24 hour periods (recall 1 and recall 2) within each method. Recall 1 and Recall 2 are in-person visits one week apart.
  Bland Altman analysis. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately.
Extent of agreement between measured and self-reported weight | The average weight in kg of the two 24 hour periods (recall 1 and recall 2) within each method. Recall 1 and Recall 2 are in-person visits one week apart.
  Bland Altman analysis. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately.
Extent of agreement between measured and self-reported height | The average height in cm of the two 24 hour periods (recall 1 and recall 2) within each method. Recall 1 and Recall 2 are in-person visits one week apart.
  Bland Altman analysis. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately.
User acceptability of the online dietary assessment tool based on the evaluation questionnaire data | At the conclusion of the second in-person visit, one week after the first in-person visit.
  Evaluation questionnaire. Data for adults, younger school age children (7-13 years) and older school age children (14-17 years) participants in different age subgroups (7-13 years, 14-17 years, 18 years and older) will be analyzed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Soshina, Study Director — PepsiCo Holdings, LLC 72/4, Leningradsky prospect, Moscow, Russian Federation, 125315
Locations (4):
- Russia (4):
  - CRO Name: OCT Rus Ltd., Saint Petersburg
  - Eco-Safety LLC, Saint Petersburg
  - Astarta, LCC, Saint Petersburg
  - Mayly LLC, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pigat S, Soshina M, Berezhnaya Y, Kryzhanovskaya E. Web-Based 24-Hour Dietary Recall Tool for Russian Adults and School-Aged Children: Validation Study. JMIR Form Res. 2023 Aug 16;7:e41774. doi: 10.2196/41774. PMID 37585243